CLINICAL TRIAL: NCT03872167
Title: Evaluation of Conventional Non-invasive Mechanical Ventilation (NIV) Versus an Automatic Ventilation Mode in Patients With NIV Criteria.
Brief Title: Evaluation of Conventional Non-invasive Mechanical Ventilation (NIV) Versus an Automatic Ventilation Mode.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, CRISTINA EMBID LOPEZ, Principal Investigator, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NIVHCLINIC
Record Dates: First submitted 2019-03-07; First posted 2019-03-13 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Hypoxemic Respiratory Failure; Hypercapnic Respiratory Failure
Keywords: NIV; hypoxemia; hypercapnia
MeSH Terms: conditions — Respiratory Insufficiency; Hypoxia; Hypercapnia | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MANUAL (Active Comparator): Manual titration of non-invasive mechanical ventilation using polysomnography and randomized
  Interventions: Device: BIPAP, manual tritration.
- AUTOMATIC (Active Comparator): Automatic titration of the non-invasive mechanical ventilation using the same device in an automatic mode with assured volume and pressure support.
  Interventions: Device: BIPAP, Intelligent automatic mode defined by assured volume with pressure support

INTERVENTIONS:
Device: BIPAP, Intelligent automatic mode defined by assured volume with pressure support — Correction of night ventilation through an automatic mode of ventilation with assured volume with pressure support
  Arms: AUTOMATIC
Device: BIPAP, manual tritration. — Correction of night ventilation through a manual titration of non-invasive mechanical ventilation using polysomnography.
  Arms: MANUAL

SUMMARY:
To evaluate the polysomnographic performance of an automatic ventilatory mode compared with the gold standard (manual polysomnographic titration) to adjust chronic non-invasive ventilation by means of a randomized cross-over study.

DETAILED DESCRIPTION:
Prospective randomized crossover study in 26 patients with chronic non-invasive ventilation (NIV) criteria, comparing the NIV titration with polysomnography vs an automatic mode of ventilation. It will be compared with clinical parameters of ventilation, blood analysis and inflammation reactants as well as evaluating the patient's comfort after each mode.

ELIGIBILITY:
Inclusion Criteria: chronic respiratory failure

* Diurnal hipercapnia and/or nocturnal hypoventilation (CT90% >10%)

Exclusion Criteria:

* Under 18 years old.
* Presence of severe uncontrolled cardiac comorbidity.
* Impossibility to achieve adaptation to therapy in the training session.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Partial pressure of carbon dioxide (PaCO2) | two weeks
  Measure levels after each polysomnography using arterial blood gases
Partial pressure of oxygen (PaO2) | two weeks
  Measure levels after each polysomnography using arterial blood gases

SECONDARY OUTCOMES:
Oxygen saving time below 90% (CT90%) | one month
  Assess the polysomnography reduction in CT90% through the night study.

CONTACTS AND LOCATIONS:
Overall Officials: CRISTINA EMBID LOPEZ, PHD, Principal Investigator — Hospital Clinic; MONICA C MATUTE VILLACIS, MD, Principal Investigator — Hospital Clinic
Locations (1):
- Hospital Clinic Barcelona., Barcelona, Spain